CLINICAL TRIAL: NCT00868621
Title: Identification of Urinary Cytokines in Patients With Overactive Bladder (OAB)
Brief Title: Urinary Cytokines in Patients With Overactive Bladder (OAB)
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB 8848
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Overactive Bladder; Urinary Tract Infection
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Control Group(CG)- Healthy age-matched volunteers with no urinary symptoms.
- 2: Overactive Bladder Patients Group(OAB)- Patients with urgency of urination.
- 3: Urinary Tract Infection Group(UTI)- Symptomatic patients with dysuria, urgency and frequency of urination with proven urine cultures of infection.

SUMMARY:
Overactive bladder (OAB) is a widespread condition characterized by urgency, urge incontinence, nocturia and excessive urinary frequency, affecting millions of people worldwide. In two epidemiological studies, OAB was found in about 17% of American and European populations. This accounts for an estimated 33 million patients suffering from OAB in the USA. The disorder constitutes a psychological stress that impacts the patient's social life.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a widespread condition characterized by urgency, urge incontinence, nocturia and excessive urinary frequency, affecting millions of people worldwide.(1) In two epidemiological studies, OAB was found in about 17% of American and European populations.(2)(3). This accounts for an estimated 33 million patients suffering from OAB in the USA. The disorder constitutes a psychological stress that impacts the patient's social life.

The luminal surface of the bladder is covered by the urothelium, which functions as a highly efficient barrier to the movement of water and ionized substances across the bladder wall.(4) Urothelial cells also have specialized sensory and signaling properties that allow them to respond to their chemical and physical environment, and engage in reciprocal chemical communication with neighboring nerves in the bladder wall. These properties are 1) nicotinic, muscarinic, tachykinin, adrenergic and capsaicin (TRPV1) receptor expression, 2) sensitivity to transmitters released from afferent and efferent nerves, 3) mechanosensitivity, 4) close physical association with afferent nerves and 5) the ability to release chemical mediators such as ATP and NO, which can regulate the activity of adjacent nerves and, thereby, trigger local vascular changes and/or reflex bladder contractions.(5)

Transmitter release from urothelial cells appears to be mediated by a calcium dependent exocytotic mechanism that is similar to the mechanism involved in transmitter release from nerve terminals. Transmitters released from urothelial cells can act in an autocrine/paracrine manner in the urothelium, or on subepithelial myofibroblasts, nerves or blood vessels to influence various functions, including the urothelial barrier, local blood flow and sensory mechanisms.(6)

Urine cytokine assays have been studied in various bladder and kidney disorders with the hope of understanding the pathophysiology and developing a noninvasive, reliable predictor of disease progression and evaluate the response to treatment.

Interstitial cystitis (IC) is a severely debilitating syndrome of unknown etiology affecting the urinary bladder that is mainly associated with urgency, frequency and pain. Pro-inflammatory molecules and neuroinflammation are suggested in the patho-mechanism of IC. Abdel Mageed and Ghoniem found out the activation of the nuclear factor kappa B (NF-k B) in the bladder biopsy of IC patients. NF-k B is a transcription factor found in some inflammatory diseases like rheumatoid arthritis, bronchial asthma, and inflammatory bowel diseases. NF-k B has a role in induction of pro inflammatory cytokines IL-6, IL-2, IL-1β and TNF-α. Activation of NF-k B was associated with 27, 8, 10 and 7 fold increase in TNF-α, IL-10, IL-6 and IL-8 transcripts respectively.(7,8) Keay et al determined that the urine of IC patients specifically contains a factor that inhibit primary bladder epithelial proliferation, anti proliferative factor (APF) and it has significantly decreased heparin binding epidermal growth factor like factor (HBEGF) and increased epidermal growth factor (EGF) levels compared to urine from normal subjects.(9) Chai et al compared urine levels of APF and HB-EGF before and after bladder distention and neurostimulation.(10,11) Both of urine markers changed toward normal levels after hydrodistention or neuromodulation treatment of IC.

Urinary cytokines have also been studied in patients undergoing intravesical bacillus Calmette Guerin (BCG) therapy for superficial bladder cancer.(12) BCG is thought to cause local immunostimulation, resulting in infiltration of T-lymphocytes in the bladder wall. After treatment, IL-1, IL-2, IL-6, and TNF are significantly elevated in the urine. It is thought that BCG induced cytokines may generate bladder tumor killing cells, and an elevation of urine cytokines may correlate clinical response to BCG therapy.

Recently, there have been studies that have attempted to identify specific measurable urinary factors that lead to the progression of chronic renal disease. Cytokines are involved in the recruitment of inflammatory cells, leading to infiltration in the diseased kidney, ultimately resulting in renal scarring. Elevated levels of urinary IL-6 and TNF receptor-1 are identified in children with vesicoureteral reflux associated with reflux nephropathy and renal scarring.(13)

Acute renal allograft rejection is a result of the recipient's immune response to the donor kidney, and 35% of these patients experience an episode of acute rejection the first year after surgery. Elevated urinary cytokines have been measured in patients who have biopsy proven renal allograft acute rejection.(14)

Urinary cytokines and markers have been identified in different urological disorders. They are used to understand the pathophysiology, diagnosis and evaluation of the treatment of these disorders. We hypothesize that there is urothelial abnormality in cases of overactive bladder that leads to elaboration of certain kinds of urinary cytokines. To our knowledge, no study has been published evaluating urinary markers in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Group I (OAB patients)

  1. Women with OAB, ≥18 years and premenopausal non-menstruating, not on any anticholinergic for at least two weeks before enrollment in the study.
  2. Significant urgency,i.e., having moderate or severe urgency score.
  3. Having a score > 8 on the OAB-V8 questionnaire.
  4. Urinary frequency of more than 8/day, with urgency of urination, with or without urge incontinence.
  5. Negative screening urinalysis one month after documented UTI.
* Group II (Control)

  1. Age-matched normal volunteers (≥18 years and premenopausal non-menstruating)
  2. No Urgency.
  3. OAB-8 score < 8.
  4. No UTI.
* Group III (UTl)

  1. Age-matched
  2. ≥18 years and premenopausal non-menstruating women with culture proven UTI.

Exclusion Criteria:

1. Treatable genitourinary conditions that could cause incontinence
2. Hematuria
3. Obstructive uropathy
4. Patients diagnosed with vaginitis
5. History of urothelial carcinoma
6. Urinary tract infection (except group III)
7. Pelvic radiation.
8. Neurogenic bladder.
9. Renal pathology.
10. Stress urinary incontinence.
11. Medications.
12. Recent history of Botox injection in the bladder (Within the last year).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty healthy women (control), 20 women suffering from overactive bladder and other 20 women suffering from UTI will be selected for the study. Each control will be age matched within +/- 5 years to patients.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Ghoniem, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Mageed AB, Bajwa A, Shenassa BB, Human L, Ghoniem GM. NF-kappaB-dependent gene expression of proinflammatory cytokines in T24 cells: possible role in interstitial cystitis. Urol Res. 2003 Oct;31(5):300-5. doi: 10.1007/s00240-003-0339-9. Epub 2003 Jul 11. PMID 14574533
- [Background] de Reijke TM, de Boer EC, Kurth KH, Schamhart DH. Urinary cytokines during intravesical bacillus Calmette-Guerin therapy for superficial bladder cancer: processing, stability and prognostic value. J Urol. 1996 Feb;155(2):477-82. PMID 8558640
- [Background] Ninan GK, Jutley RS, Eremin O. Urinary cytokines as markers of reflux nephropathy. J Urol. 1999 Nov;162(5):1739-42. PMID 10524926
- [Background] Lewis SA. Everything you wanted to know about the bladder epithelium but were afraid to ask. Am J Physiol Renal Physiol. 2000 Jun;278(6):F867-74. doi: 10.1152/ajprenal.2000.278.6.F867. PMID 10836974
- [Background] Chopra B, Barrick SR, Meyers S, Beckel JM, Zeidel ML, Ford AP, de Groat WC, Birder LA. Expression and function of bradykinin B1 and B2 receptors in normal and inflamed rat urinary bladder urothelium. J Physiol. 2005 Feb 1;562(Pt 3):859-71. doi: 10.1113/jphysiol.2004.071159. Epub 2004 Dec 2. PMID 15576455
- [Background] Kanai A, de Groat W, Birder L, Chai T, Hultgren S, Fowler C, Fry C. Symposium report on urothelial dysfunction: pathophysiology and novel therapies. J Urol. 2006 May;175(5):1624-9. doi: 10.1016/S0022-5347(05)00977-8. PMID 16600715
- [Background] Kim JC, Park EY, Seo SI, Park YH, Hwang TK. Nerve growth factor and prostaglandins in the urine of female patients with overactive bladder. J Urol. 2006 May;175(5):1773-6; discussion 1776. doi: 10.1016/S0022-5347(05)00992-4. PMID 16600756
- [Background] Yokoyama O, Yusup A, Miwa Y, Oyama N, Aoki Y, Akino H. Effects of tolterodine on an overactive bladder depend on suppression of C-fiber bladder afferent activity in rats. J Urol. 2005 Nov;174(5):2032-6. doi: 10.1097/01.ju.0000176793.50410.9e. PMID 16217388
- [Background] Yokoyama O, Yusup A, Oyama N, Aoki Y, Tanase K, Matsuta Y, Miwa Y, Akino H. Improvement of bladder storage function by alpha1-blocker depends on the suppression of C-fiber afferent activity in rats. Neurourol Urodyn. 2006;25(5):461-7. doi: 10.1002/nau.20253. PMID 16673377
- [Background] Thongboonkerd V, McLeish KR, Arthur JM, Klein JB. Proteomic analysis of normal human urinary proteins isolated by acetone precipitation or ultracentrifugation. Kidney Int. 2002 Oct;62(4):1461-9. doi: 10.1111/j.1523-1755.2002.kid565.x. PMID 12234320
- [Background] Townsend JC, Sadler WA, Shanks GM. The effect of storage pH on the precipitation of proteins in deep frozen urine samples. Ann Clin Biochem. 1987 Jan;24 ( Pt 1):111-2. doi: 10.1177/000456328702400118. No abstract available. PMID 3827174
- [Background] Tadros Y, Ruiz-Deya G, Crawford BE, Thomas R, Abdel-Mageed AB. In vivo proteomic analysis of cytokine expression in laser capture-microdissected urothelial cells of obstructed ureteropelvic junction procured by laparoscopic dismembered pyeloplasty. J Endourol. 2003 Jun;17(5):333-6. doi: 10.1089/089277903322145530. PMID 12885361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Urine samples from Patients with Uninary Track Infection(UTI)and OAB attending Cleveland Clinic Florida (CCF) clinics were entered after screening).
  Urine samples were collected from age-matched Volunteers.
Pre-assignment Details: Aliquots of urine were centrifuged, frozen and stored at -80 degrees celcius. Samples were shipped on dry ice to co-authors by overnight courier. Co-authors were blinded to which samples were OAB, control or UTI.
Groups:
- Normal Patients - Control: Healthy age-matched volunteers with no urinary symptoms
- Overactive Bladder Patients: Patients urgency if urination
- Urinary Tract Infection: Symptomatic patients with dysuria, urgency and frequency of urination with proven urine cultures of infection.
Period: Overall Study
Arm/Group | Normal Patients - Control | Overactive Bladder Patients | Urinary Tract Infection
Started | 20 | 20 | 20
Completed | 20 | 20 | 16 (16 patients included and 4 patients had negative urine cultures, and were excluded)
Not Completed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Patients - Control | Overactive Bladder Patients | Urinary Tract Infection | Total
Number analyzed (Participants) | 20 | 20 | 16 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 16 | 56
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (4.5) | 29 (5) | 26.5 (6) | 27.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 16 | 56
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 16 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elevated Cytokines (Levels of Pro-inflammatory)
Description: Used commercial human cytokine chip. If the study proved that certain cytokines are significantly present (p<0.05 compared to a standard) in the urine of OAB patients, further research to study the effect of anticholinergic drugs on the level of these cytokines in urine will be conducted.
Time Frame: 18 months
Population: Normal Patients - Control:Urine analysis showing no UTI Overactive Bladder Patients: Urgency of urination, but negative UTI Urinary Tract Infection: Symptoms + Positive urine culture
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Patients - Control | Overactive Bladder Patients | Urinary Tract Infection
Number analyzed (Participants) | 20 | 20 | 16
Participants | 20 | 20 | 16

ADVERSE EVENTS:
Description: There were "0" adverse events since no subject intervention was done. Test was performed only on voided urine samples and Adverse Events were not collected or observed.
Arm/Group | Normal Patients - Control | Overactive Bladder Patients | Urinary Tract Infection
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small numbers of participants, results need to be verified by other methods (quantitative)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No